CLINICAL TRIAL: NCT05292625
Title: Outcomes of Umbilical Cord -derived Mesenchymal Stem Cell Infusion in Patients with Neurological Sequelae After Ischemic Stroke
Brief Title: Stem Cell Infusion in the Treatment of Patients with Neurological Sequelae After Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VinmecISC1809
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; umbilical cord mesenchymal stem cells; Neurological Complication
MeSH Terms: conditions — Ischemic Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- UC-MSC infusion via intravenous route (Experimental): 1.5 x 10^6 umbilical Cord Mesenchymal Stem Cells per body kg will be infusion via the intravenous at baseline, and the second transplantation will be performed 3 months after the first transplantation and combination with standard frailty treatment and supplementary medication
  Interventions: Biological: UC-MSC infusion via intravenous route; Other: standard stroke treatment and rehabilitation therapy
- UC-MSC infusion via intrathecal route (Experimental): 1.5 x 10^6 umbilical Cord Mesenchymal Stem Cells per body kg will be infusion via the intrathecal at baseline, and the second transplantation will be performed 3 months after the first transplantation and combination with standard frailty treatment and supplementary medication
  Interventions: Biological: UC-MSC infusion via intrathecal route; Other: standard stroke treatment and rehabilitation therapy
- control arm (Other): standard stroke treatment and rehabilitation therapy
  Interventions: Other: standard stroke treatment and rehabilitation therapy

INTERVENTIONS:
Biological: UC-MSC infusion via intravenous route — Patients assigned to UC-MSC administration groups will receive two administrations at a dose of 1.5 million cells/kg patient body weight via the intravenous (IV) route with a 3-month intervening interval
  Arms: UC-MSC infusion via intravenous route
Biological: UC-MSC infusion via intrathecal route — Patients assigned to UC-MSC administration groups will receive two administrations at a dose of 1.5 million cells/kg patient body weight via the intrathecal route with a 3-month intervening interval
  Arms: UC-MSC infusion via intrathecal route
Other: standard stroke treatment and rehabilitation therapy — Each patient can receive up to 30 days of rehabilitation therapy

SUMMARY:
This trial is to investigate the safety and potential therapeutic efficacy of allogeneic administration of umbilical cord-derived MSCs (UC-MSCs) in combination with standard neurological complications after ischemic stroke treatment in Vietnam.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death behind ischemic heart disease worldwide. Traditional treatments have some limitations whereas preclinical data suggest that stem cell therapy is a promising regenerative medical treatment given the limited capacity of the central nervous system for self-repairs after ischemic stroke. Previous studies have shown that umbilical cord blood-derived Mesenchymal stem cell (UC-MSC) infusion improves the outcomes of several neurological damage conditions, including stroke. These results encouraged us to initiate the phase I/II clinical trial aiming to evaluate the safety and the efficiency of UC-MSC transplantation in the treatment of patients with neurological complications after ischemic stroke. This case-control phase I/II trial is conducted at Vinmec Times City International Hospital, Hanoi, Vietnam between 2021 and 2023. In this trial, 48 patients with neurological complications after ischemic stroke will be enrolled into 3 groups: UC-MSC infusion via intravenous route group (16), UC-MSC infusion via intrathecal administration route group (16), and control group (16). The UC-MSC group (IV/intrathecal) will receive two doses of thawed UC-MSC product at 1.5x106 cells/kg patient body weight with an intervention interval of three months. The primary outcome measures will include the incidence of prespecified administration-associated adverse events (AEs) and serious adverse events (SAEs). The potential efficacy will be measured using these scales including National Institutes of Health Stroke Scale-NIHSS, Functional Independence Measure -FIM, Modified Ashworth Scale-MAS, Fine motor skills-FMS, 36-Item Short Form Survey -SF-36. The clinical evaluation will be conducted at baseline and 3-, 6- and 12-months post-intervention.

ELIGIBILITY:
* Age: from 40 to 75 years.
* Gender: either sex
* Patients have been discharged/patients who are hospitalized but their general condition is stable:

  * No need for vasopressor drugs
  * No need for mechanical ventilation or oxygen support
  * No signs of infection (fever, high WBC, high CRP/Procalcitonin)
  * No kidney failure, liver failure, heart failure.
* Time from onset to study participation ≤ 24 months
* National Institutes of Health Stroke Scale (NIHSS) score >=5
* Agree to participate in the study

Exclusion Criteria:

* Hematologic cause of stroke
* There is evidence of active infections, failure of heart, lung, liver, or kidney, respiratory distress syndrome, anemia, clotting disorder
* Cancer.
* Pregnancy.
* Tracheostomy, coma, complete quadriplegia, vegetative.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | up to the 12-month period following treatment
  To assess safety, the number of AEs or SAEs during stem cell administration (72 h) at 3 months, 6 months and 12 months after discharge will be evaluated

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) score | up to the 12-month period following treatment
  National Institutes of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating more severe neurological deficit
Functional Independence Measure (FIM) score | up to the 12-month period following treatment
  Functional Independence Measure (FIM) is a widely accepted functional assessment measure used during inpatient rehabilitation with the possible total score ranging from 18 (lowest) to 126 (highest) level of independence
Modified Ashworth Scale | up to the 12-month period following treatment
  The modified Ashworth scale purpose is to grade muscle spasticity. The scale is from 0 (No increase in muscle tone) to 4 (affected part(s) rigid in flexion or extension)
Fine motor skills (FMI) score | up to the 12-month period following treatment
  Fine motor skills (FMI) scores range from 0 to 58
Short Form 36 items (SF-36) score | up to the 12-month period following treatment
  Short Form 36 items (SF-36) consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability

CONTACTS AND LOCATIONS:
Overall Officials: Liem T Nguyen, Prof, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen LT, Nguyen TTN, Nguyen KT, Phung LN, Hoang VT, Phan TTK, Van Pham M, Nguyen ATP, Van Ngo D, Van Nguyen A, Van Nguyen C. Intrathecal versus intravenous umbilical cord mesenchymal stem cells for ischemic stroke sequelae. Stem Cells Transl Med. 2025 Nov 24;14(12):szaf063. doi: 10.1093/stcltm/szaf063. PMID 41277536
- [Derived] Hoang VT, Le DS, Hoang DM, Phan TTK, Ngo LAT, Nguyen TK, Bui VA, Nguyen Thanh L. Impact of tissue factor expression and administration routes on thrombosis development induced by mesenchymal stem/stromal cell infusions: re-evaluating the dogma. Stem Cell Res Ther. 2024 Feb 27;15(1):56. doi: 10.1186/s13287-023-03582-3. PMID 38414067